CLINICAL TRIAL: NCT07235371
Title: Transcutaneous Electrical Acupoint Stimulation on Postoperative Urinary Retention After Radical Surgery for Cervical Cancer: A Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation for Postoperative Urinary Retention After Radical Surgery for Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lu Chao (Other)
Responsible Party: Sponsor-Investigator, Lu Chao, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2025-1262
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Urinary Retention (POUR)
Keywords: Postoperative urinary retention,; POUR; TEAS; transcutaneous electrical acupoint stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The TEAS Group (Experimental): Participants will receive TEAS treatment once a day for two consecutive weeks. TEAS stimulation: A set of TEAS patch stimulation will be applied to BL32 and BL34 points on both sides of the spine respectively, with an intensity of approximately 30 ± 5mA, based on patient tolerance. The frequency will be 2/10Hz.
  Interventions: Other: transcutaneous electrical acupoint stimulation
- The Sham TEAS Group (Placebo Comparator): Participants will receive sham TEAS treatment once a day for two consecutive weeks. The operation of the sham TEA group will be consistent with that of the TEAS group, with a current intensity set to 30mA. However, the instrument circuit of the fake TEAS group cannot output current normally, and participants can only feel patches stimulating at the BL32 and BL34 acupoints.
  Interventions: Other: Sham transcutaneous electrical acupoint stimulation

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation — Participants will receive TEAS treatment once a day for two consecutive weeks. TEAS stimulation: A set of TEAS patch stimulation will be applied to BL32 and BL34 points on both sides of the spine respectively, with an intensity of approximately 30 ± 5mA, based on patient tolerance. The frequency will be 2/10Hz.
  Other Names: TEAS
  Arms: The TEAS Group
Other: Sham transcutaneous electrical acupoint stimulation — Participants will receive sham TEAS treatment once a day for two consecutive weeks. The operation of the sham TEAS group will be consistent with that of the TEAS group, with a current intensity set at 30 mA. However, the instrument circuit of the fake TEAS group cannot output current normally, and participants can only feel patches stimulating at the BL32 and BL34 acupoints.
  Other Names: Sham TEAS
  Arms: The Sham TEAS Group

SUMMARY:
This is a prospective, blinded, single-center, randomized controlled trial. We will include 76 patients with postoperative urinary retention (POUR) after radical hysterectomy for cervical cancer who have a clear diagnosis and meet the screening criteria as the research object. They will be randomly divided into the transcutaneous electrical acupoint stimulation（TEAS）group and the sham TEAS group according to a 1:1 ratio. Each group consists of 38 patients, and all patients will be required to sign a written informed consent form. The TEAS group will be treated with TEAS based on conventional treatment, and the sham TEAS group will be treated with shamTEAS based on conventional treatment. The main outcomes will be the changes in post-void residual (PVR) volume; secondary indicators will include the response rate of participants with successful urinary catheter removal after intervention, assessment of urinary tract infection (UTI), and patient quality of life assessment according to the EORTC QLQ-C30 scale. The participants will also be evaluated with expectations, blind evaluation, compliance evaluation, and safety evaluation to preliminarily evaluate the effect of TEAS for postoperative urinary retention after radical hysterectomy for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age range of 18-70 years, expected survival period ≥ 6 months; (2) Meets diagnostic criteria, with an indwelling catheter duration of more than 14 days but less than 1 year; (3) No history of urinary system diseases before surgery; (4) Clear consciousness, unobstructed communication, daily living ability, patients or family members can learn TEAS operation; (5) No serious systemic diseases such as heart, liver, brain, kidney, etc; (6) Karnofsky functional status score (KPS) ≥ 70 points; (7) Voluntarily participate and sign a written informed consent form.

Exclusion Criteria:

* (1) Obstructive urinary retention, such as urethral stricture or stones; (2) combined with other serious systemic diseases, advanced cachexia; (3) Patients with pacemaker implantation or metal implantation in the body; (4) The treatment site has skin lesions or is not suitable for TEAS treatment in other populations; (5) Physical or mental disorders with cognitive impairment; (6) Other clinical trial participants who are currently involved in affecting the results of this study; (7) Those who do not agree to participate in clinical trials; (8) The evaluator has determined that the participant is not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
The change in post-void residual (PVR) volume of the bladder | week 2 (after intervention), and week 4 （follow-up）
  It will use a direct measurement method to detect residual urine volume in the bladder.

SECONDARY OUTCOMES:
The response rate of participants who will successfully remove the urinary catheter | week 2 （after intervention）
  The participants in each group who will remove their urinary catheters after intervention (week 2), in proportion to the total number of patients in each group, multiplied by 100%. It can also be understood as the initial cure rate of POUR.
The proportion of patients who have a urinary tract infection (UTI). | Week 0 (baseline), week 2 (after intervention), and week 4 （follow-up）
  Determine whether the patient has a urinary tract infection based on their urine routine test or urine culture test results.
The evaluation of the quality of life | week 0 (baseline), week 2 (after intervention), and week 4 （follow-up）
  Assessing patients' quality of life using the EQRTC QLQ-C30 scale.
Safety Assessment | week 2 （after intervention）, and week 4 (follow-up)
  Evaluate based on the Adverse Event Scale.

OTHER OUTCOMES:
Participant Expectation Value Evaluation | week 0 (baseline)
  Evaluate based on the participant's expected value scale
Blinding evaluation | week 2（after intervention）
  Evaluate according to the established blind assessment questionnaire
Participant compliance assessment | week 2 （after intervention）and week 4（follow-up）
  Evaluate based on the participant compliance assessment scale

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No